CLINICAL TRIAL: NCT05482568
Title: Phase IB/II Clinical Study of the Safety, Tolerability, Pharmacokinetics, and Efficacy of Injectable SHR-A1811 in Combination With Pyrotinib or SHR-1316 in Subjects With Advanced Non-small Cell Lung Cancer With HER2
Brief Title: A Trial of Injectable SHR-A1811 in Combination With Pyrotinib or SHR-1316 in Subjects With Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-II-203
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Intervention Model Description: An open, multicenter, dose-increasing/investigational Phase IB/II clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 combined with Pyrotinib/SHR-A1811 combined with SHR-1316 (Experimental)
  Interventions: Drug: SHR-A1811 & Pyrotinib/SHR-A1811 & SHR-1316

INTERVENTIONS:
Drug: SHR-A1811 & Pyrotinib/SHR-A1811 & SHR-1316 — Drug: SHR-A1811 & Pyrotinib
  SHR-A1811： intravenous Pyrotinib：oral
  Drug: SHR-A1811 & SHR-1316
  SHR-A1811： intravenous SHR-1316： intravenous

SUMMARY:
This study was an open, multicenter, dose-increasing/investigational Phase IB/II clinical trial to evaluate the efficacy of SHR-A1811 in combination with other antitumor therapies in subjects with advanced non-small cell lung cancer with HER2 . It can be divided into two parts, Part A is the dose escalation and efficacy exploration study of SHR-A1811 combined with Pyrotinib, and Part B is the dose escalation and efficacy exploration study of SHR-A1811 combined with SHR-1316.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent, signed and dated IRB/EC approved informed consent, willing and able to comply with treatment planning visits, tests and other procedural requirements
2. When signing the informed consent, the age is 18-75 years old (including both ends), and there is no gender limitation
3. The ECOG score is 0 or 1
4. The expected survival is ≥12 weeks
5. Subjects with advanced or metastatic non-small cell lung cancer
6. Formalin fixed, paraffin-embedded tumor tissue blocks or sections of unstained tumor specimens are provided
7. Subjects who have failed prior standard care or are intolerant to standard care
8. There is at least one measurable lesion
9. Vital organs are functioning well
10. Heart function is good
11. Agree to birth control

Exclusion Criteria:

1. There are untreated or active central nervous system (CNS) tumor metastases
2. Pleural, ascites, or pericardial effusion requiring intervention occurred within 7 days prior to initial administration
3. Systemic antitumor therapy was performed 4 weeks prior to study initiation
4. Prior treatment with antibody-conjugated drugs
5. Received >30 Gy chest radiation within 6 months prior to initial administration
6. Palliative radiotherapy was completed within 7 days prior to initial administration
7. Failure to recover from toxicity and/or complications of previous interventions to nCI-CTCAE ≤1
8. The half-life of CYP3A4 suppressor, moderate inhibitor or strong inducer or moderate inducer is less than 3 or less than 14 days from the date of first drug use, and the shorter is selected
9. Received systemic immunosuppressant therapy within 14 days prior to the first study
10. Subjects with known or suspected interstitial pneumonia
11. In the first study, failure to swallow, chronic diarrhea, gastroenteritis, intestinal obstruction, gastrointestinal perforation, postgastrectomy, or colitis, or other medical conditions or special conditions affecting drug administration and absorption occurred within 28 days prior to administration
12. Presence of any active, known or suspected autoimmune disease
13. Have poorly controlled or severe cardiovascular disease
14. Previous or concurrent malignancy
15. Subjects who developed a severe infection within 28 days prior to the first dose
16. Active hepatitis B
17. There were active tuberculosis patients within 1 year before enrollment
18. There is a history of immunodeficiency
19. Live attenuated vaccine was administered within 28 days prior to initial study administration or is expected to be administered during study treatment
20. Subjects who are participating in another clinical study or who have had their first dose less than 4 weeks since the end of the previous clinical study (last dose) or 5 half-lives of the study drug, whichever is shorter
21. Major surgery other than diagnosis or biopsy was performed within 28 days prior to initial administration
22. People who are known to be allergic to sir-A1811, pyrrolitinib, or any of the components of SIR-1316
23. History of severe allergic reactions to other monoclonal antibody/fusion protein drugs
24. Female subjects who are pregnant, breast-feeding, or planning to become pregnant during the study
25. Uncontrolled mental illness and other conditions known to affect the completion of the study process, such as alcohol, drug or substance abuse and detention
26. Any other conditions that, in the investigator's judgment, may increase the risk of study participation, interfere with study results, or make study participation unsuitable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
DLT(Phase I (dose exploration phase) main study endpoint) | 21 days after the first administration of each subject
AE(Phase I (dose exploration phase) main study endpoint) | Two years after the last subject was enrolled in the group
Incidence and severity of serious adverse events (SAE)(Phase I (dose exploration phase) main study endpoint) | Two years after the last subject was enrolled in the group
Objective response rate(The main end points of the second stage (efficacy expansion stage)) | Two years after the last subject was enrolled in the group

SECONDARY OUTCOMES:
Toxin binding antibody to shr-a1811（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Total antibody to shr-a1811（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Plasma concentration of free toxin shr169265（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Plasma concentration of pyrroltinib（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Plasma concentration of SHR-1316（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Anti shr-a1811 antibody positive（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
The positive status of neutralizing antibody against shr-a1811（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Anti shr-1316 antibody positive（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
The positive status of neutralizing antibody against shr-1316（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Objective Response Rate（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Duration of response（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
Progression Free Survival（Phase I secondary endpoint） | Two years after the last subject was enrolled in the group
AE（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Incidence and severity of serious adverse events (SAE)（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Toxin binding antibody to shr-a1811（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Total antibody to shr-a1811（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Plasma concentration of free toxin shr169265（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Plasma concentration of pyrroltinib（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Plasma concentration of SHR-1316（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Anti shr-a1811 antibody positive（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
The positive status of neutralizing antibody against shr-a1811（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Anti shr-1316 antibody positive（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
The positive status of neutralizing antibody against shr-1316（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Duration of response（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group
Progression Free Survival（Phase II secondary study endpoint） | Two years after the last subject was enrolled in the group

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Chest hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided